CLINICAL TRIAL: NCT00518336
Title: Follow-up Study to Evaluate the Long-term Efficacy of a HPV Vaccine (580299) in Healthy Young Adult Women in Brazil
Brief Title: Follow-up Study to Evaluate the Long-term Efficacy of the HPV Vaccine (580299) in Healthy Young Adult Women in Brazil
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 109616 (Y7); 109624 (Other: GSK); 109625 (Other: GSK)
Record Dates: First submitted 2007-08-17; First posted 2007-08-20 (Estimated); Results first posted 2011-10-25 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-10

CONDITIONS: Infections, Papillomavirus
MeSH Terms: conditions — Papillomavirus Infections | interventions — Blood Specimen Collection; human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Cervarix Group (Experimental): Young adult women from the Brazilian cohort who participated in the primary study 580299/001 (NCT00689741) and follow-up study 580299/007 (NCT00120848) and received 3 doses of Cervarix at 0, 1 and 6 months intramuscularly into the deltoid region of the non-dominant arm during the primary study.
  Interventions: Procedure: Blood sampling; Procedure: Collection of cervical specimen; Biological: Cervarix
- Placebo Group (Placebo Comparator): Young adult women from the Brazilian cohort who participated in the primary study 580299/001 (NCT00689741) and follow-up study 580299/007 (NCT00120848) and received 3 doses of placebo at 0, 1 and 6 months intramuscularly into the deltoid region of the non-dominant arm during the primary study.
  Interventions: Procedure: Blood sampling; Procedure: Collection of cervical specimen

INTERVENTIONS:
Procedure: Blood sampling — Blood sampling at Visit 3, 5 and 7.
Procedure: Collection of cervical specimen — Collection of cervical specimen at Visit2, 3, 4, 5, 6 and 7.
Biological: Cervarix — Three doses administered intramuscularly at 0, 1 and 6 months.
  Arms: Cervarix Group

SUMMARY:
Infection with human papillomavirus (HPV) has been clearly established as the central cause of cervical cancer. This Phase IIb study is designed to evaluate the the long-term efficacy, safety and immunogenicity of the 580299 HPV vaccine (CervarixTM) in a Brazilian cohort of women vaccinated in the phase IIb, blinded, primary study 580299/001 (NCT00689741) and having participated in follow-up study 580299/007 (NCT00120848). Only subjects who participated in the primary & follow-up study will be enrolled in this long-term follow-up study. Subjects were aged 15-25 years at the time of entry into the primary study.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
In this extension study, women who were vaccinated in the primary study, and participated in the follow-up study, will be followed with visits every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* Subjects who participated in study 580299-007.
* Written informed consent obtained from the subject prior to enrollment.

Exclusion Criteria:

* Use or planned use of any investigational or non-registered product other than the study vaccine.
* Decoding of the subject's 580299-001 treatment allocation to either the subject or the investigator.
* Administration or planned administration of any other HPV vaccine, other than the vaccine administered in study 580299-001.

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 433 (Actual)
Dates: Start 2007-11; Primary Completion 2008-07 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Brazil (5):
  - GSK Investigational Site, Curitiba, Paraná
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, São Paulo, São Paulo
  - GSK Investigational Site, Campinas
  - GSK Investigational Site, Fortaleza

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Naud PS, Roteli-Martins CM, De Carvalho NS, Teixeira JC, de Borba PC, Sanchez N, Zahaf T, Catteau G, Geeraerts B, Descamps D. Sustained efficacy, immunogenicity, and safety of the HPV-16/18 AS04-adjuvanted vaccine: final analysis of a long-term follow-up study up to 9.4 years post-vaccination. Hum Vaccin Immunother. 2014;10(8):2147-62. doi: 10.4161/hv.29532. PMID 25424918
- [Derived] Roteli-Martins CM, Naud P, De Borba P, Teixeira JC, De Carvalho NS, Zahaf T, Sanchez N, Geeraerts B, Descamps D. Sustained immunogenicity and efficacy of the HPV-16/18 AS04-adjuvanted vaccine: up to 8.4 years of follow-up. Hum Vaccin Immunother. 2012 Mar;8(3):390-7. doi: 10.4161/hv.18865. Epub 2012 Feb 13. PMID 22327492
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 109616 (Y7) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109616 (Y7) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 109616 (Y7) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 109624 are summarised with studies 109616 and 109625 on the GSK Clinical Study Register.
- Available data/document: Informed Consent Form: 109616 (Y7) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109616 (Y7) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109616 (Y7) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the five subjects withdraw at Year 7, three subjects came back during Year 8 and are therefore not longer considered as withdraw subjects. At Year 9, one subject, who did not participate to Year 7 and Year 8 visits, came back for one of the visits and was added to Total cohort.
Period: Year 7
Arm/Group | Cervarix Group | Placebo Group
Started | 222 | 211
Completed | 220 | 208
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Could not attend in time | 0 | 3
Period: Year 8
Arm/Group | Cervarix Group | Placebo Group
Started | 223 (1 subject withdrawn at Year 7 came back and was therefore no longer considered as withdrawn.) | 213 (2 subjects withdrawn at Year 7 came back and were therefore no longer considered as withdrawn.)
Completed | 222 | 211
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Could not attend in time | 0 | 1
Period: Year 9
Arm/Group | Cervarix Group | Placebo Group
Started | 224 (1 subject did not particpate at the previous timepoint, came back and was added in the Total cohort) | 213
Completed | 219 | 212
Not Completed | 5 | 1
Not completed — Migrated/moved from study area | 1 | 1
Not completed — Lost to Follow-up | 3 | 0
Not completed — Personal reasons | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix Group | Placebo Group | Total
Number analyzed (Participants) | 222 | 211 | 433
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (3.2) | 26.4 (2.9) | 26.5 (3.05)
Gender [Count of Participants; unit: Participants]
  Female | 222 | 211 | 433
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Presenting Cervical Infections With Human Papillomavirus (HPV) -16 and/or HPV-18
Description: Cervical HPV infection was defined as the first detection of an HPV type in a subject previously negative for that HPV type.
Time Frame: Up to year 8
Population: According-To-Protocol (ATP) cohort for analysis of efficacy included all subjects for whom differential treatment effect on efficacy was likely (i.e. who met all eligibility criteria in the primary study (580299/001), the first follow-up (580299/007) and the current study), who complied with the protocol and for whom efficacy data were available.
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 178 | 139
subjects
  HPV-16 (N=176;122) | 0 | 5
  HPV-18 (N=178;133) | 0 | 4
  HPV-16/18 (N=176;139) | 0 | 5

2. Secondary Outcome: Number of Subjects Presenting Cervical Infections With Any Oncogenic HPV Type
Description: Oncogenic HPV types included HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
  Subjects with an event did not report the same event in the earlier studies. Subjects were DNA negative for the 14 oncogenic HPV types and had a normal cytology at baseline in the primary study. Subjects with an event were DNA negative for the corresponding HPV type at month 6 in the primary study.
Time Frame: Up to year 8
Population: The ATP cohort for analysis of efficacy included all subjects for whom differential treatment effect on efficacy was likely (i.e. who met all eligibility criteria in the primary study (580299/001), the first follow-up (580299/007) and the current study), who complied with the protocol and for whom efficacy data were available.
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 154 | 135
subjects
  Including HPV-16 or 18 (N=154; 133) | 32 | 39
  Without HPV-16 or 18 (N=154; 135) | 32 | 36

3. Secondary Outcome: Number of Subjects Presenting Cervical Infections With Individual Oncogenic Non-vaccine HPV Type
Description: Oncogenic types included HPV-31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
  Subjects with an event did not report the same event in the earlier studies and were DNA negative for the corresponding HPV type at month 6 in the primary study.
Time Frame: Up to year 8
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 201 | 180
subjects
  HPV-31 (N=195; 168) | 1 | 5
  HPV-33 (N=195; 175) | 0 | 1
  HPV-35 (N=195; 177) | 4 | 5
  HPV-39 (N=189; 162) | 4 | 2
  HPV-45 (N=201; 174) | 3 | 5
  HPV-51 (N=166; 152) | 4 | 10
  HPV-52 (N=170; 152) | 15 | 9
  HPV-56 (N=181; 168) | 2 | 4
  HPV-58 (N=189; 173) | 4 | 2
  HPV-59 (N=193; 180) | 2 | 1
  HPV-66 (N= 176; 164) | 3 | 8
  HPV-68 (N= 186; 166) | 6 | 6

4. Secondary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With HPV-16 and/or HPV-18
Description: Persistent cervical HPV infection (6-month definition) was defined as detection of the same HPV type in cervical specimens at 2 consecutive evaluations over a minimum of 5 months.
  Subjects with an event did not report the same event in the earlier studies. Subjects were DNA negative for the 14 oncogenic HPV types and had a normal cytology at baseline in the primary study. Subjects with an event were DNA negative for the corresponding HPV type at month 6 in the primary study.
Time Frame: Up to year 8
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 178 | 151
subjects
  HPV-16/18 (N=178; 144) | 0 | 0
  HPV-16 (N=178; 149) | 0 | 0
  HPV-18 (N=178;151) | 0 | 0

5. Secondary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With Any Oncogenic HPV Types
Description: Oncogenic HPV types included HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
  Persistent cervical HPV infection (6-month definition) was defined as detection of the same HPV type in cervical specimens at 2 consecutive evaluations over a minimum of 5 months.
  Subjects with an event did not report the same event in the earlier studies. Subjects were DNA negative for the 14 oncogenic HPV types and had a normal cytology at baseline in the primary study. Subjects with an event were DNA negative for the corresponding HPV type at month 6 in the primary study.
Time Frame: Up to year 8
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 162 | 143
subjects
  Including HPV-16 or 18 (N=162; 142) | 15 | 17
  Without HPV-16 or 18 (N=162; 143) | 15 | 17

6. Secondary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With Individual Oncogenic Non-vaccine HPV Types
Description: Oncogenic HPV types included HPV-31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
  Persistent cervical HPV infection (6-month definition) was defined as detection of the same HPV type in cervical specimens at 2 consecutive evaluations over a minimum of 5 months.
  Subjects with an event did not report the same event during the earlier studies. Subjects with an event were DNA negative for the corresponding HPV type at Month 6 in the primary study.
Time Frame: Up to year 8
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 203 | 184
Subjects
  HPV-31 (N= 201; 180) | 1 | 4
  HPV-33 (N= 199; 182) | 1 | 1
  HPV-35 (N= 200; 180) | 2 | 3
  HPV-39 (N= 199; 174) | 2 | 2
  HPV-45 (N= 203; 184) | 4 | 1
  HPV-51 (N= 191; 174) | 3 | 3
  HPV-52 (N= 185; 166) | 4 | 4
  HPV-56 (N= 196; 182) | 1 | 2
  HPV-58 (N= 195; 181) | 3 | 3
  HPV-59 (N=202; 184) | 0 | 0
  HPV-66 (N= 191; 171) | 1 | 2
  HPV-68 (N= 199; 181) | 2 | 2

7. Secondary Outcome: Number of Subjects With Persistent Infection (12-month Definition) With HPV-16 and/or HPV-18
Description: Persistent cervical HPV infection (12-month definition) was defined as detection of the same HPV type in cervical specimens at all consecutive evaluations over a minimum of 10 months.
  Subjects with an event did not report the same event in the earlier studies. Subjects were DNA negative for the 14 oncogenic HPV types and had a normal cytology at baseline in the primary study. Subjects with an event were DNA negative for the corresponding HPV type at month 6 in the primary study.
Time Frame: Up to year 8
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 178 | 156
subjects
  HPV-16/18 (N= 178; 152) | 0 | 0
  HPV-16 (N= 178; 154) | 0 | 0
  HPV-18 (N= 178; 156) | 0 | 0

8. Secondary Outcome: Number of Subjects With Persistent Infection (12-month Definition) With Any Oncogenic HPV Types
Description: Oncogenic HPV types included HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
  Persistent cervical HPV infection (12-month definition) was defined as detection of the same HPV type in cervical specimens at all consecutive evaluations over a minimum of 10 months.
  Subjects with an event did not report the same event in the earlier studies. Subjects were DNA negative for the 14 oncogenic HPV types and had a normal cytology at baseline in the primary study. Subjects with an event were DNA negative for the corresponding HPV type at month 6 in the primary study.
Time Frame: Up to year 8
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 163 | 143
subjects
  Including HPV-16 or 18 (N= 163; 142) | 8 | 3
  Without HPV-16 or 18 (N= 163; 143) | 8 | 3

9. Secondary Outcome: Number of Subjects With Persistent Infection (12-month Definition) With Individual Oncogenic Non-vaccine HPV Types
Description: Individual oncogenic non-vaccine HPV types include HPV-31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
  Persistent cervical HPV infection (12-month definition) was defined as detection of the same HPV type in cervical specimens at all consecutive evaluations over a minimum of 10 months.
  Subjects with an event did not report the same event in the earlier studies and were DNA negative for the corresponding HPV type at month 6 in the primary study.
Time Frame: Up to year 8
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 204 | 186
subjects
  HPV-31 (N= 202; 181) | 1 | 2
  HPV-33 (N= 202; 184) | 1 | 0
  HPV-35 (N= 200; 185) | 0 | 1
  HPV- 39 (N= 200; 179) | 2 | 1
  HPV-45 (N= 204; 186) | 3 | 1
  HPV- 51 (N= 198; 182) | 1 | 1
  HPV-52 (N= 191; 172) | 3 | 1
  HPV-56 (N= 200; 185) | 0 | 0
  HPV-58 (N= 199; 183) | 0 | 1
  HPV-59 (N= 203; 186) | 0 | 0
  HPV-66 (N= 195; 177) | 0 | 1
  HPV-68 (N= 200; 184) | 1 | 0

10. Secondary Outcome: Number of Subjects With Histopathologically-confirmed Cervical Intraepithelial Neoplasia (CIN)1+ Associated With HPV-16 or HPV-18 Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: CIN1+ was defined as CIN (Cervical Intraepithelial Neoplasia) grades 1,2 and 3, adenocarcinoma in situ (AIS) and invasive cervical cancer.
  Subjects with an event did not report the same event in the earlier studies. Subjects were DNA negative for the 14 oncogenic HPV types and had normal cytology at baseline in the primary study. Subjects with an event were DNA negative for the corresponding HPV type at Month 6 in the primary study.
Time Frame: Up to year 8
Population: The analysis was performed on the Total Cohort, which included all enrolled subjects who came at the first visit and received at least one vaccine dose (Cervarix or placebo)
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 199 | 186
subjects
  HPV-16/18 (N= 199; 182) | 0 | 0
  HPV-16 (N= 199; 183) | 0 | 0
  HPV-18 (N= 199; 186) | 0 | 0

11. Secondary Outcome: Number of Subjects With Histopathologically Confirmed CIN1+ Associated With Oncogenic HPV Types Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: CIN1+ was defined as CIN grades 1,2 and 3, adenocarcinoma in situ (AIS) and invasive cervical cancer.
  Oncogenic HPV types assessed included HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
  Subjects with an event did not report the same event in the earlier studies. Subjects were DNA negative for the 14 oncogenic HPV types and had normal cytology at baseline in the primary study. Subjects with an event were DNA negative for the corresponding HPV type at Month 6 in the primary study.
Time Frame: Up to year 8
Population: as for outcome 10
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 199 | 187
subjects
  Including HRV-16 or 18 | 0 | 1
  Without HRV-16 or 18 | 0 | 1

12. Secondary Outcome: Number of Subjects With Histopathologically Confirmed CIN1+ Associated With Individual Oncogenic Non-Vaccine HPV Types Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: CIN1+ was defined as CIN grades 1,2 and 3, adenocarcinoma in situ (AIS) and invasive cervical cancer.
  Oncogenic HPV types assessed included HPV-31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
  Subjects with an event did not report the same event in the earlier studies and were DNA negative for the corresponding HPV type at Month 6 in the primary study.
Time Frame: Up to year 8
Population: as for outcome 10
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 222 | 209
subjects
  HPV-31 (N= 221; 207) | 0 | 0
  HPV-33 (N= 220; 207) | 0 | 0
  HPV-35 (N= 219; 206) | 0 | 0
  HPV-39 (N= 222; 209) | 0 | 0
  HPV-45 (N= 221; 208) | 0 | 0
  HPV-51 (N= 215; 206) | 0 | 0
  HPV-52 (N= 218; 204) | 0 | 1
  HPV-56 (N= 219; 209) | 0 | 1
  HPV-58 (N=221; 206) | 0 | 0
  HPV-59 (N=220; 208) | 0 | 0
  HPV-66 (N= 219; 203) | 0 | 0
  HPV-68 (N= 221; 209) | 0 | 0

13. Secondary Outcome: Number of Subjects With Histopathologically-confirmed CIN2+ Associated With HPV-16 or HPV-18 Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: CIN2+ was defined as CIN grades 2 and 3, AIS and invasive cervical cancer.
  Subjects with an event did not report the same event in the earlier studies. Subjects were DNA negative for the 14 oncogenic HPV types and had normal cytology at baseline in the primary study. Subjects with an event were DNA negative for the corresponding HPV type at Month 6 in the primary study.
Time Frame: Up to year 8
Population: as for outcome 10
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 199 | 186
subjects
  HPV-16/18 (N= 199; 184) | 0 | 0
  HPV-16 (N= 199; 185) | 0 | 0
  HPV-18 (N= 199; 186) | 0 | 0

14. Secondary Outcome: Number of Subjects With Histopathologically Confirmed CIN2+ Associated With Oncogenic HPV Types Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: CIN2+ was defined as CIN grades 2 and 3, AIS and invasive cervical cancer.
  Oncogenic HPV types assessed included HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
  Subjects with an event did not report the same event in the earlier studies. Subjects were DNA negative for the 14 oncogenic HPV types and had normal cytology at baseline in the primary study. Subjects with an event were DNA negative for the corresponding HPV type at Month 6 in the primary study.
Time Frame: Up to year 8
Population: as for outcome 10
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 199 | 187
subjects
  Including HPV-16 or 18 | 0 | 0
  Without HPV-16 or 18 | 0 | 0

15. Secondary Outcome: Number of Subjects With Histopathologically Confirmed CIN2+ Associated With Individual Oncogenic Non-Vaccine HPV Types Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: CIN2+ was defined as CIN grades 2 and 3, AIS and invasive cervical cancer.
  Oncogenic HPV types assessed included HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
  Subjects with an event did not report the same event in the earlier studies. and were DNA negative for the corresponding HPV type at Month 6 in the primary study.
Time Frame: Up to year 8
Population: as for outcome 10
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 222 | 209
subjects
  HPV-31 (N= 221; 208) | 0 | 0
  HPV-33 (N= 220; 208) | 0 | 0
  HPV-35 (N= 220; 206) | 0 | 0
  HPV-39 (N= 222; 209) | 0 | 0
  HPV-45 (N= 221; 208) | 0 | 0
  HPV-51 (N= 217; 207) | 0 | 0
  HPV-52 (N= 218; 206) | 0 | 1
  HPV-56 (N= 219; 209) | 0 | 0
  HPV-58 (N= 221; 207) | 0 | 0
  HPV-59 (N= 220; 208) | 0 | 0
  HPV-66 (N= 220; 205) | 0 | 0
  HPV-68 (N= 221; 209) | 0 | 0

16. Secondary Outcome: Number of Subjects With Abnormal Cytology Greater Than or Equal to Atypical Squamous Cells of Undetermined Significance (ASC-US) Associated With an HPV 16 and/or HPV-18 Cervical Infection
Description: Abnormal cytology included atypical squamus cells of undetermined significance (ASC-US), low-grade squamous intraepithelial lesion (LSIL), high-grade squamous intraepithelial lesion (HSIL), atypical glandular cells (AGC), atypical squamus cells and cannot exclude HSIL (ASC-H).
  Subjects with an event did not report the same event in the earlier studies. Subjects were DNA negative for the 14 oncogenic HPV types and had normal cytology at baseline in the primary study. Subjects with an event were DNA negative for the corresponding HPV type at Month 6 in the primary study.
Time Frame: Up to year 8
Population: as for outcome 10
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 199 | 177
subjects
  HPV-16/18 (N= 198; 165) | 0 | 1
  HPV-16 (N= 198; 171) | 0 | 0
  HPV-18 (N= 199; 177) | 0 | 1

17. Secondary Outcome: Number of Subjects With Abnormal Cytology Greater Than or Equal to Atypical Squamous Cells of Undetermined Significance (ASC-US) Associated With Oncogenic HPV Types Cervical Infection
Description: Abnormal cytology included ASC-US, LSIL, HSIL, AGC, and ASC-H.
  Oncogenic HPV types assessed included HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
  Subjects with an event did not report the same event in the earlier studies. Subjects were DNA negative for the 14 oncogenic HPV types and had normal cytology at baseline in the primary study. Subjects with an event were DNA negative for the corresponding HPV type at Month 6 in the primary study.
Time Frame: Up to year 8
Population: as for outcome 10
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 196 | 184
subjects
  Including HPV-16 or 18 (N= 196; 183) | 10 | 15
  Without HPV-16 or 18 (N= 196; 184) | 10 | 15

18. Secondary Outcome: Number of Subjects With Abnormal Cytology Greater Than or Equal to Atypical Squamous Cells of Undetermined Significance (ASC-US) Associated With Individual Oncogenic Non-vaccine HPV Types Cervical Infection
Description: Abnormal cytology included ASC-US, LSIL, HSIL, AGC and ASC-H.
  Oncogenic HPV types assessed included HPV-31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
  Subjects with an event did not report the same event in the earlier studies and were DNA negative for the corresponding HPV type at month 6 in the primary study.
Time Frame: Up to year 8
Population: as for outcome 10
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 220 | 206
subjects
  HPV-31 (N= 217; 200) | 0 | 5
  HPV-33 (N= 218; 202) | 0 | 1
  HPV-35 (N= 217; 202) | 1 | 1
  HPV-39 (N= 217; 197) | 1 | 1
  HPV-45 (N= 220; 204) | 2 | 0
  HPV-51 (N= 202; 194) | 1 | 3
  HPV-52 (N= 205; 183) | 3 | 3
  HPV-56 (N= 207; 202) | 1 | 1
  HPV-58 (N= 213; 199) | 0 | 3
  HPV-59 (N= 216; 206) | 0 | 1
  HPV-66 (N= 214; 194) | 2 | 1
  HPV-68 (N= 217; 202) | 2 | 1

19. Secondary Outcome: Number of Subjects With Abnormal Cytology Greater Than or Equal to Low-grade Squamous Intraepithelial Lesion (LSIL) Associated With an HPV 16 and/or HPV-18 Cervical Infection
Description: Abnormal cytology included ASC-US, LSIL, HSIL, AGC and ASC-H.
  Subjects with an event did not report the same event in the earlier studies. Subjects were DNA negative for the 14 oncogenic HPV types and had normal cytology at baseline in the primary study. Subjects with an event were DNA negative for the corresponding HPV type at Month 6 in the primary study.
Time Frame: Up to year 8
Population: as for outcome 10
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 199 | 183
subjects
  HPV-16/18 (N= 198; 174) | 0 | 1
  HPV-16 (N= 198; 177) | 0 | 0
  HPV-18 (N= 199; 183) | 0 | 1

20. Secondary Outcome: Number of Subjects With Abnormal Cytology Greater Than or Equal to Low-grade Squamous Intraepithelial Lesion (LSIL) Associated With Oncogenic HPV Types Cervical Infection
Description: as for outcome 17
Time Frame: Up to year 8
Population: as for outcome 10
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 197 | 186
subjects
  Including HPV-16 or 18 | 7 | 12
  Without HPV-16 or 18 | 7 | 12

21. Secondary Outcome: Number of Subjects With Abnormal Cytology Greater Than or Equal to Low-grade Squamous Intraepithelial Lesion (LSIL) Associated With Individual Oncogenic Non-vaccine HPV Types Cervical Infection
Description: as for outcome 18
Time Frame: Up to year 8
Population: as for outcome 10
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 220 | 207
subjects
  HPV-31 (N= 218; 202) | 0 | 4
  HPV-33 (N= 219; 205) | 0 | 1
  HPV-35 (N= 217; 204) | 0 | 0
  HPV-39 (N= 219; 200) | 1 | 1
  HPV-45 (N= 220; 205) | 2 | 0
  HPV-51 (N= 211; 197) | 1 | 3
  HPV-52 (N= 210; 191) | 2 | 3
  HPV-56 (N= 211; 202) | 1 | 0
  HPV-58 (N= 216; 203) | 0 | 2
  HPV-59 (N= 219; 207) | 0 | 1
  HPV-66 (N= 217; 195) | 0 | 1
  HPV-68 (N= 219; 206) | 2 | 1

22. Secondary Outcome: Anti-HPV-16 and Anti-HPV-18 Enzyme-linked Immunosorbent Assay (ELISA) Titers in the Immunogenicity Cohort
Description: Titers are given as Geometric Mean Titers (GMTs) expressed as ELISA Units per milliliter (EL.U/mL).
Time Frame: At Months 77-101
Population: The analyses were performed on the ATP cohort for immunogenicity, which included evaluable subjects for whom immunogenicity data were available.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 111 | 68
EL.U/mL
  Anti-HPV-16 Month 77-82 (N= 69; 54) | 374.9 [291.8 to 481.8] | 5.4 [4.4 to 6.6]
  Anti-HPV-16 Month 83-88 (N= 111; 68) | 383.4 [312.9 to 469.9] | 5.1 [4.4 to 6.0]
  Anti-HPV-16 Month 89-94 (N= 94; 67) | 346.3 [270.3 to 443.6] | 5.4 [4.4 to 6.7]
  Anti-HPV-16 Month 95-101 (N= 87; 56) | 435.1 [347.5 to 544.9] | 5.4 [4.4 to 6.6]
  Anti-HPV-18 Month 77-82 (N= 69; 54) | 252.8 [196.9 to 324.7] | 4.3 [3.7 to 5.1]
  Anti-HPV-18 Month 83-88 (N= 111; 68) | 251.0 [208.7 to 301.8] | 5.0 [4.1 to 6.1]
  Anti-HPV-18 Month 89-94 (N= 94; 67) | 234.6 [188.8 to 291.5] | 4.4 [3.7 to 5.2]
  Anti-HPV-18 Month 95-101 (N= 87; 56) | 246.5 [197.6 to 307.5] | 4.6 [3.7 to 5.6]

23. Secondary Outcome: Anti-HPV-16 and Anti-HPV-18 Pseudovirion-based Neutralization Assay (PBNA) Titers in the Immunogenicity Subset
Description: Data are expressed as Geometric Mean Titers (GMTs). The titer is the serum dilution giving a 50 percent reduction of the signal compared to a control without serum
Time Frame: At Months 77-101
Population: The analyses were performed on a subset of the ATP cohort for immunogenicity, which included evaluable subjects for whom immunogenicity data were available.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 30 | 8
titer
  Anti-HPV-16 Month 77-82 (N= 15; 4) | 1616.1 [592.7 to 4407.0] | 20.0 [20.0 to 20.0]
  Anti-HPV-16 Month 83-88 (N= 30; 8) | 1990.7 [1228.5 to 3225.8] | 20.0 [20.0 to 20.0]
  Anti-HPV-16 Month 89-94 (N= 18; 6) | 1385.0 [740.6 to 2590.0] | 20.0 [20.0 to 20.0]
  Anti-HPV-16 Month 95-101 (N= 27; 6) | 1611.6 [934.1 to 2780.3] | 20.0 [20.0 to 20.0]
  Anti-HPV-18 Month 77-82 (N= 15; 4) | 845.4 [361.6 to 1976.7] | 20.0 [20.0 to 20.0]
  Anti-HPV-18 Month 83-88 (N= 30; 8) | 751.6 [466.3 to 1211.5] | 20.0 [20.0 to 20.0]
  Anti-HPV-18 Month 89-94 (N= 18; 6) | 1185.3 [656.1 to 2141.1] | 20.0 [20.0 to 20.0]
  Anti-HPV-18 Month 95-101 (N= 27; 6) | 578.2 [352.9 to 947.1] | 20.0 [20.0 to 20.0]

24. Secondary Outcome: Number of Subjects With New Onset Chronic Diseases (NOCD) up to Year 7
Description: NOCDs include for example asthma, type I diabetes, allergies, ...
Time Frame: Up to year 7
Population: as for outcome 10
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 222 | 211
subjects | 0 | 0

25. Secondary Outcome: Number of Subjects With NOCD up to Year 8
Description: NOCDs included for example asthma, type I diabetes, allergies, ...
  NOCDs which were not unblinded at the subject level at the time of the analysis are not presented and will be disclosed as soon as they become available.
Time Frame: Up to year 8
Population: as for outcome 10
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 223 | 213
subjects | 5 | 2

26. Secondary Outcome: Number of Subjects With New Onset Autoimmune Disease (NOAD) up to Year 7
Time Frame: Up to year 7
Population: as for outcome 10
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 222 | 211
subjects | 0 | 0

27. Secondary Outcome: Number of Subjects With NOAD up to Year 8
Description: The values of NOADs are not yet corresponding to the values in each group. The cases are still blinded. They will be disclosed as soon as the results will be available.
Time Frame: Up to year 8
Population: as for outcome 10
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 223 | 213
subjects | 2 | 2

28. Secondary Outcome: Number of Subjects With Medically Significant Conditions up to Year 7
Description: Medically significant conditions include adverse events (AEs) prompting emergency room or physician visits that are not related to common diseases or routine visits for physical examination or vaccination, or serious adverse events (SAEs) that are not related to common diseases. Common diseases include upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervico-vaginal yeast infections, menstrual cycle abnormalities and injury.
  Medically significant conditions which were not unblinded at the time of the analysis are not presented yet.
Time Frame: Up to year 7
Population: as for outcome 10
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 222 | 211
subjects | 18 | 13

29. Secondary Outcome: Number of Subjects With Medically Significant Conditions up to Year 8
Description: as for outcome 28
Time Frame: up to year 8
Population: as for outcome 10
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 223 | 213
subjects | 40 | 24

30. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) up to Year 7
Description: SAEs assessed include medical occurrences that result in death, is life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject
Time Frame: Up to year 7
Population: as for outcome 10
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 222 | 211
subjects | 4 | 5

31. Secondary Outcome: Number of Subjects With SAEs up to Year 8
Description: as for outcome 30
Time Frame: up to year 8
Population: as for outcome 10
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 223 | 213
subjects | 10 | 7

32. Secondary Outcome: Number of Subjects Presenting Cervical Infections With Any Oncogenic HPV Type.
Description: as for outcome 2
Time Frame: Up to year 9
Population: The According -To-Protocol (ATP) cohort for efficacy included all subjects for whom differential treatment effect on efficacy was likely (i.e. those meeting all eligibility criteria in the primary study (580299/001), the first follow-up (580299/007) and the current study), who complied with the protocol and for whom efficacy data were available.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 155 | 136
Subjects
  Including HPV-16 or 18 (N=155;135) | 38 | 49
  Without HPV-16 or 18 (N=155;136) | 38 | 45

33. Secondary Outcome: Number of Subjects Presenting Cervical Infections With Individual Oncogenic Non-vaccine HPV Type
Description: as for outcome 3
Time Frame: Up to year 9
Population: as for outcome 32
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 203 | 182
Subjects
  HPV-31 (N=197;170) | 4 | 5
  HPV-33 (N=197;177) | 2 | 4
  HPV-35 (N=197;179) | 4 | 9
  HPV-39 (N=191;163) | 5 | 3
  HPV-45 (N=203;176) | 3 | 5
  HPV-51 (N=167;154) | 11 | 15
  HPV-52 (N=172;153) | 18 | 10
  HPV-56 (N=182;170) | 3 | 4
  HPV-58 (N=191;175) | 7 | 3
  HPV-59 (N=195;182) | 2 | 2
  HPV-66 (N=176;165) | 4 | 10
  HPV-68 (N=188;166) | 8 | 9

34. Secondary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With HPV-16 and/or HPV-18
Description: as for outcome 4
Time Frame: Up to year 9
Population: The According -To-Protocol (ATP) cohort for efficacy included all subjects for whom differential treatment effect on efficacy was likely (i.e. those meeting all eligibility criteria in the primary study (580299/001), the first follow-up (580299/007) and the current study, who complied with the protocol and for whom efficacy data were available.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 179 | 152
Subjects
  HPV-16/18 (N=179;144) | 0 | 4
  HPV-16 (N=179;149) | 0 | 3
  HPV-18 (N=179;152) | 0 | 3

35. Secondary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With Any Oncogenic HPV Type
Description: as for outcome 5
Time Frame: Up to year 9
Population: The According-To-Protocol (ATP) cohort for efficacy included all subjects for whom differential treatment effect on efficacy was likely (i.e. those meeting all eligibility criteria in the primary study (580299/001), the first follow-up (580299/007) and the current study), who complied with the protocol and for whom efficacy data were available.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 163 | 144
Subjects
  Including HPV-16 or 18 (N=163;143) | 20 | 25
  Without HPV-16 or 18 (N=163;144) | 20 | 24

36. Secondary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With Individual Oncogenic Non-vaccine HPV Types
Description: as for outcome 6
Time Frame: Up to year 9
Population: as for outcome 35
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 205 | 186
Subjects
  HPV-31 (N=203;182) | 1 | 4
  HPV-33 (N=201;184) | 1 | 1
  HPV-35 (N=202;182) | 4 | 4
  HPV-39 (N=201;176) | 3 | 2
  HPV-45 (N=205;186) | 4 | 1
  HPV-51 (N=193;176) | 4 | 4
  HPV-52 (N=187;167) | 6 | 7
  HPV-56 (N=198;184) | 1 | 3
  HPV-58 (N=197;183) | 5 | 3
  HPV-59 (N=204;186) | 0 | 1
  HPV-66 (N=192;172) | 1 | 5
  HPV-68 (N=201;182) | 4 | 2

37. Secondary Outcome: Number of Subjects With Persistent Infection (12-month Definition) With HPV-16 and/or HPV-18
Description: as for outcome 7
Time Frame: Up to year 9
Population: as for outcome 35
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 179 | 157
Subjects
  HPV-16/18 (N=179;153) | 0 | 1
  HPV-16 (N=179;155) | 0 | 0
  HPV-18 (N=179;157) | 0 | 2

38. Secondary Outcome: Number of Subjects With Persistent Infection (12-month Definition) With Any Oncogenic HPV Types
Description: as for outcome 8
Time Frame: Up to year 9
Population: as for outcome 35
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 164 | 144
Subjects
  Including HPV-16 or 18 (N=164;143) | 13 | 10
  Without HPV-16 or 18 (N=164;144) | 13 | 8

39. Secondary Outcome: Number of Subjects With Persistent Infection (12-month Definition) With Individual Oncogenic Non-vaccine HPV Types
Description: as for outcome 9
Time Frame: Up to year 9
Population: as for outcome 35
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 206 | 188
Subjects
  HPV-31 (N=204,183) | 1 | 4
  HPV-33 (N=204;186) | 1 | 0
  HPV-35 (N=202;187) | 2 | 2
  HPV-39 (N=202;181) | 2 | 1
  HPV-45 (N=206;188) | 4 | 1
  HPV-51 (N=200;184) | 2 | 2
  HPV-52 (N=193;174) | 3 | 3
  HPV-56 (N=202;187) | 0 | 0
  HPV-58 (N=201;185) | 1 | 1
  HPV-59 (N=205;188) | 0 | 0
  HPV-66 (N=196;179) | 0 | 1
  HPV-68 (N=202;185) | 2 | 0

40. Secondary Outcome: Number of Subjects With Histopathologically-confirmed CIN1+ Associated With HPV-16 or HPV-18 Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: Cervical Intraepithelial Neoplasia (CIN1)+ was defined as CIN grades 1,2 and 3, adenocarcinoma in situ (AIS) and invasive cervical cancer.
  Subjects with an event did not report the same event in the earlier studies. Subjects were DNA negative for the 14 oncogenic HPV types and had normal cytology at baseline in the primary study. Subjects with an event were DNA negative for the corresponding HPV type at Month 6 in the primary study.
Time Frame: Up to year 9
Population: The analyses was performed on the Total Cohort, which included all enrolled subjects who came at the first visit and received at least one vaccine dose (Cervarix or Placebo)
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 200 | 187
Subjects
  HPV-16/18 (N=200;183) | 0 | 1
  HPV-16 (N=200;184) | 0 | 1
  HPV-18 (N=200;187) | 0 | 0

41. Secondary Outcome: Number of Subjects With Histopathologically Confirmed CIN1+ Associated With Oncogenic HPV Types Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: as for outcome 11
Time Frame: Up to year 9
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 200 | 188
Subjects
  Including HPV-16 or 18 (N=200;188) | 3 | 4
  Without HPV-16 or 18 (N=200;188) | 3 | 4

42. Secondary Outcome: Number of Subjects With Histopathologically Confirmed CIN1+ Associated With Individual Oncogenic Non-Vaccine HPV Types Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: as for outcome 12
Time Frame: Up to year 9
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 224 | 211
Subjects
  HPV-31 (N=223;209) | 0 | 1
  HPV-33 (N=222;209) | 0 | 0
  HPV-35 (N=221;208) | 1 | 0
  HPV-39 (N=224;211) | 0 | 0
  HPV-45 (N=223;210) | 0 | 0
  HPV-51 (N=217;208) | 0 | 0
  HPV-52 (N=220;206) | 2 | 2
  HPV-56 (N=221;211) | 0 | 1
  HPV-58 (N=223;208) | 0 | 2
  HPV-59 (N=222;210) | 0 | 1
  HPV-66 (N=220;205) | 0 | 0
  HPV-68 (N=223;210) | 2 | 0

43. Secondary Outcome: Number of Subjects With Histopathologically-confirmed CIN2+ Associated With HPV-16 or HPV-18 Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: as for outcome 13
Time Frame: Up to year 9
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 200 | 187
Subjects
  HPV-16/18 (N=200;185) | 0 | 0
  HPV-16 (N=200;186) | 0 | 0
  HPV-18 (N=200;187) | 0 | 0

44. Secondary Outcome: Number of Subjects With Histopathologically Confirmed CIN2+ Associated With Oncogenic HPV Types Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: as for outcome 14
Time Frame: Up to year 9
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 200 | 188
Subjects
  Including HPV-16 or 18 (N=200;188) | 0 | 2
  Without HPV-16 or 18 (N=200;188) | 0 | 2

45. Secondary Outcome: Number of Subjects With Histopathologically Confirmed CIN2+ Associated With Individual Oncogenic Non-Vaccine HPV Types Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: CIN2+ was defined as CIN grades 2 and 3, AIS and invasive cervical cancer.
  Oncogenic HPV types assessed included HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
  Subjects with an event did not report the same event in the earlier studies and were DNA negative for the corresponding HPV type at Month 6 in the primary study.
Time Frame: Up to year 9
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 224 | 211
Subjects
  HPV-31 (N=223;210) | 0 | 1
  HPV-33 (N=222;210) | 0 | 0
  HPV-35 (N=222;208) | 0 | 0
  HPV-39 (N=224;211) | 0 | 0
  HPV-45 (N=223;210) | 0 | 0
  HPV-51 (N=219;209) | 0 | 0
  HPV-52 (N=220;208) | 0 | 1
  HPV-56 (N=221;211) | 0 | 0
  HPV-58 (N=223;209) | 0 | 2
  HPV-59 (N=222;210) | 0 | 0
  HPV-66 (N=221;207) | 0 | 0
  HPV-68 (N=223;210) | 0 | 0

46. Secondary Outcome: Number of Subjects With Abnormal Cytology Greater Than or Equal to Atypical Squamous Cells of Undertermined Significance (ASC-US) Associated With an HPV 16 and/or HPV-18 Cervical Infection
Description: as for outcome 16
Time Frame: Up to year 9
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 200 | 178
Subjects
  HPV-16/18 (N=199;165) | 0 | 3
  HPV-16 (N=199;171) | 0 | 1
  HPV-18 (N=200;178) | 0 | 2

47. Secondary Outcome: Number of Subjects With Abnormal Cytology Greater Than or Equal to Atypical Squamous Cells of Undertermined Significance (ASC-US) Associated With Oncogenic HPV Types Cervical Infection
Description: as for outcome 17
Time Frame: Up to year 9
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 197 | 185
Subjects
  Including HPV-16 or 18 (N=197;184) | 15 | 25
  Without HPV-16 or 18 (N=197;185) | 15 | 25

48. Secondary Outcome: Number of Subjects With Abnormal Cytology Greater Than or Equal to Atypical Squamous Cells of Undertermined Significance (ASC-US) Associated With Individual Oncogenic Non-vaccine HPV Types Cervical Infection
Description: as for outcome 18
Time Frame: Up to year 9
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 222 | 208
Subjects
  HPV-31 (N=219;202) | 1 | 5
  HPV-33 (N=220;204) | 0 | 2
  HPV-35 (N=219;204) | 1 | 3
  HPV-39 (N=219;198) | 1 | 1
  HPV-45 (N=222;206) | 2 | 0
  HPV-51 (N=203;196) | 3 | 7
  HPV-52 (N=207;184) | 5 | 5
  HPV-56 (N=208;204) | 1 | 1
  HPV-58 (N=215;201) | 3 | 4
  HPV-59 (N=218;208) | 0 | 2
  HPV-66 (N=214;195) | 2 | 2
  HPV-68 (N=219;202) | 2 | 2

49. Secondary Outcome: Number of Subjects With Abnormal Cytology Greater Than or Equal to Low-grade Squamous Intraepithelial Lesion (LSIL) Associated With an HPV 16 and/or HPV-18 Cervical Infection
Description: as for outcome 19
Time Frame: Up to year 9
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 200 | 184
Subjects
  HPV-16/18 (N=199;174) | 0 | 2
  HPV-16 (N=199;177) | 0 | 1
  HPV-18 (N=200;184) | 0 | 1

50. Secondary Outcome: Number of Subjects With Abnormal Cytology Greater Than or Equal to Low-grade Squamous Intraepithelial Lesion (LSIL) Associated With Oncogenic HPV Types Cervical Infection
Description: as for outcome 17
Time Frame: Up to year 9
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 198 | 187
Subjects
  Including HPV-16 or 18 (N=198;187) | 12 | 19
  Without HPV-16 or 18 (N=198;187) | 12 | 19

51. Secondary Outcome: Number of Subjects With Abnormal Cytology Greater Than or Equal to Low-grade Squamous Intraepithelial Lesion (LSIL) Associated With Individual Oncogenic Non-vaccine HPV Types Cervical Infection
Description: as for outcome 18
Time Frame: Up to year 9
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 222 | 209
Subjects
  HPV-031 (N=220;204) | 1 | 5
  HPV-33 (N=221;207) | 0 | 2
  HPV-35 (N=219;206) | 0 | 0
  HPV-39 (N=221;201) | 1 | 1
  HPV-45 (N=222;207) | 2 | 0
  HPV-51 (N=212;199) | 2 | 5
  HPV-52 (N=212;192) | 4 | 5
  HPV-56 (N=212;204) | 1 | 0
  HPV-58 (N=218;205) | 2 | 3
  HPV-59 (N=221;209) | 0 | 1
  HPV-66 (N=217;196) | 0 | 2
  HPV-68 (N=221;206) | 2 | 1

52. Secondary Outcome: Anti-HPV-16 and Anti-HPV-18 Enzyme-linked Immunosorbent Assay (ELISA) Titers in the Immunogenicity Cohort
Description: Titers are given as Geometric Mean Titers (GMTs) expressed as Enzyme-linked immunosorbent assay (ELISA) Units per milliliter (EL.U/mL).
  The cut-off-vales assessed were >= 8 or 7 EL. U/mL for anti-HPV-16 and 18, respectively.
Time Frame: At Month 77 until year 9 (Month 113)
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: EL. U/mL
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 111 | 65
EL. U/mL
  Anti-HPV-16 Month 77-82 (N=69;52) | 374.9 [291.8 to 481.8] | 5.2 [4.3 to 6.2]
  Anti-HPV-16 Month 83-88 (N=111;65) | 383.4 [312.9 to 469.9] | 5.2 [4.4 to 6.1]
  Anti-HPV-16 Month 89-94 (N=94;65) | 346.3 [270.3 to 443.6] | 5.4 [4.4 to 6.7]
  Anti-HPV-16 Month 95-100 (N=87;53) | 435.1 [347.5 to 544.9] | 5.4 [4.4 to 6.7]
  Anti-HPV-16 Month 101-106 (N=87;63) | 322.8 [249.4 to 417.6] | 5.2 [4.3 to 6.3]
  Anti-HPV-16 Month 107-113 (N=92;60) | 418.3 [344.0 to 508.6] | 6.1 [4.9 to 7.8]
  Anti-HPV-18 Month 77-82 (N=69;52) | 252.8 [196.9 to 324.7] | 4.2 [3.6 to 4.9]
  Anti-HPV-18 Month 83-88 (N=111;65) | 251.0 [208.7 to 301.8] | 5.0 [4.1 to 6.1]
  Anti-HPV-18 Month 89-94 (N=94;65) | 234.6 [188.8 to 291.5] | 4.4 [3.7 to 5.2]
  Anti-HPV-18 Month 95-100 (N=87;53) | 246.5 [197.6 to 307.5] | 4.6 [3.7 to 5.8]
  Anto-HPV-18 Month 101-106 (N=87;63) | 225.0 [177.1 to 285.8] | 4.1 [3.6 to 4.6]
  Anti-HPV-18 Month 107-113 (N=92;60) | 242.6 [199.3 to 295.2] | 4.8 [3.9 to 6.0]

53. Secondary Outcome: Anti-HPV-16 and Anti-HPV-18 Pseudovirion-based Neutralization Assay (PBNA) Titers in the Immunogenicity Subset
Description: as for outcome 23
Time Frame: At Month 77 until year 9 (Month 113)
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 30 | 8
Titer
  Anti-HPV-16 Month 77-82 (N=15;4) | 1616.1 [592.7 to 4407.0] | 20.0 [20.0 to 20.0]
  Anti-HPV-16 Month 83-88 (N=30;8) | 1990.7 [1228.5 to 3225.8] | 20.0 [20.0 to 20.0]
  Anti-HPV-16 Month 89-94 (N=18;6) | 1385.0 [740.6 to 2590.0] | 20.0 [20.0 to 20.0]
  Anti-HPV-16 Month 95-101 (N=27;6) | 1611.6 [934.1 to 2780.3] | 20.0 [20.0 to 20.0]
  Anti-HPV-16 Month 101-106 (N=16;7) | 1380.7 [667.5 to 2855.8] | 20.0 [20.0 to 20.0]
  Anti-HPV-16 Month 107-113 (N=30;5) | 1549.8 [1027.9 to 2336.8] | 20.0 [20.0 to 20.0]
  Anti-HPV-18 Month 77-82 (N=15;4) | 845.4 [361.6 to 1976.7] | 20.0 [20.0 to 20.0]
  Anti-HPV-18 Month 83-88 (N=30;8) | 751.6 [466.3 to 1211.5] | 20.0 [20.0 to 20.0]
  Anti-HPV-18 Month 89-94 (N=18;6) | 1185.3 [656.1 to 2141.1] | 20.0 [20.0 to 20.0]
  Anti-HPV-18 Month 95-101 (N=27;6) | 578.2 [352.9 to 947.1] | 20.0 [20.0 to 20.0]
  Anti-HPV-18 Month 101-106 (N=16;7) | 860.1 [441.0 to 1677.3] | 20.0 [20.0 to 20.0]
  Anti-HPV-18 Month 107-113 (N=30;5) | 552.0 [358.5 to 850.1] | 20.0 [20.0 to 20.0]

54. Secondary Outcome: Number of Subjects With New Onset Chronic Diseases (NOCD) up to Year 9
Description: NOCDs include for example asthma, type I diabetes, allergies, ...
Time Frame: Up to year 9
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 224 | 213
Subjects
  Number of Subjects With NOCD up to Year 9 | 6 | 3
  Hypothyroidism | 2 | 1
  Drug hypersensitivity | 1 | 0
  Rhinitis allergic | 0 | 1
  Type 2 diabetes mellitus | 1 | 0
  Rheumatoid arthritis | 1 | 0
  Dermatitis allergic | 0 | 1
  Skin reaction | 1 | 0
  Vitiligo | 1 | 0
  Hypertension | 1 | 0

55. Secondary Outcome: Number of Subjects With New Onset Autoimmune Disease (NOAD) up to Year 9.
Time Frame: Up to year 9
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 224 | 213
Subjects
  Number of Subjects With NOAD up to Year 9 | 4 | 1
  Hypothyroidism | 2 | 1
  Rheumatoid arthritis | 1 | 0
  Vitiligo | 1 | 0

56. Secondary Outcome: Number of Subjects With Medically Signifant Conditions up to Year 9
Description: Medically significant conditions include adverse events (AEs) prompting emergency room or physician visits that are not related to common diseases or routine visits for physical examination or vaccination, or serious adverse events (SAEs) that are not related to common diseases. Common diseases include upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervico-vaginal yeast infections, menstrual cycle abnormalities and injury.
Time Frame: Up to year 9
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 224 | 213
Subjects
  Medically Signifant Conditions up to Year 9 | 60 | 38
  Gastritis | 5 | 2
  Hypertension | 5 | 2
  Abortion spontaneous incomplete | 5 | 1
  Depression | 5 | 1
  Nephrolithiasis | 3 | 0
  Abortion missed | 2 | 2
  Hypothyroidism | 2 | 1
  Panic disorder | 2 | 1
  Bursitis | 2 | 0
  Ovarian cyst | 2 | 0
  Ovarian disorder | 2 | 0
  Anaemia | 0 | 2
  Gynaecological chlamydia infection | 0 | 2
  Pneumonia | 0 | 1
  Pyelonephritis | 0 | 1
  Blood pressure increased | 0 | 1
  Bipolar disorder | 0 | 1
  Genital herpes | 0 | 3
  Haemorrhoids | 0 | 1
  Peptic ulcer | 0 | 1
  Vomiting | 0 | 1
  Chest pain | 0 | 1
  Cholelithiasis | 0 | 1
  Breast infection | 0 | 1
  Dengue fever | 0 | 1
  Erysipelas | 0 | 1
  Gingival abscess | 0 | 1
  Pelvic inflammatory disease | 0 | 1
  Staphylococcal infection | 0 | 1
  Toxoplasmosis | 0 | 1
  Abnormal loss of weight | 0 | 1
  Metabolic syndrome | 0 | 1
  Cervical spinal stenosis | 0 | 1
  Synovial cyst | 0 | 1
  Tendonitis | 0 | 1
  Benign breast neoplasm | 0 | 1
  Benign hydatidiform mole | 0 | 1
  Ovarian cancer | 0 | 1
  Headache | 0 | 1
  Blighted ovum | 0 | 1
  Intra-uterine death | 0 | 1
  Oligohydramnios | 0 | 1
  Pre-eclampsia | 0 | 1
  Rhinitis allergic | 0 | 1
  Dermatitis allergic | 0 | 1
  Sexual abuse | 0 | 1
  Haematoma | 0 | 1

57. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) up to Year 9.
Description: as for outcome 30
Time Frame: up to year 9
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 224 | 213
Subjects | 20 | 11

58. Primary Outcome: Number of Subjects Presenting Cervical Infections With Human Papillomavirus (HPV) -16 and/or HPV-18
Description: as for outcome 1
Time Frame: Up to year 9
Population: as for outcome 35
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 179 | 140
Subjects
  HPV-16 (N=179;133) | 0 | 9
  HPV-18 (N=177;140) | 0 | 6
  HPV-16/18 (N=177;122) | 0 | 9

59. Primary Outcome: Number of Subjects Presenting Cervical Infections With Human Papillomavirus (HPV) -16 and /or HPV-18
Description: as for outcome 1
Time Frame: Up to year 7
Population: as for outcome 32
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 171 | 133
Subjects
  HPV-16 (N=171;128) | 0 | 2
  HPV-18 (N=169;133) | 0 | 0
  HPV-16/18 (N=169;117) | 0 | 2

60. Secondary Outcome: Number of Subjects Presenting Cervical Infections With Any Oncogenic HPV Type.
Description: as for outcome 2
Time Frame: Up to year 7
Population: as for outcome 32
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 148 | 126
Subjects
  Including HPV-16 or 18 (N=148;122) | 22 | 16
  Without HPV-16 or 18 (N=148;126) | 22 | 14

61. Secondary Outcome: Number of Subjects Presenting Cervical Infections With Individual Oncogenic Non-vaccine HPV Type.
Description: as for outcome 3
Time Frame: Up to year 7
Population: as for outcome 32
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 193 | 174
Subjects
  HPV-31 (N=187;162) | 1 | 1
  HPV-33 (N=187;168) | 0 | 1
  HPV-35 (N=187;170) | 3 | 3
  HPV-39 (N=181;156) | 2 | 0
  HPV-45 (N=193;167) | 2 | 3
  HPV-51 (N=158;146) | 2 | 3
  HPV-52 (N=162;147) | 10 | 3
  HPV-56 (N=174;162) | 0 | 0
  HPV-58 (N=182;166) | 2 | 0
  HPV-59 (N=186;174) | 1 | 0
  HPV-66 (N=169;157) | 3 | 3
  HPV-68 (N=179;159) | 4 | 2

62. Secondary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With HPV-16 and/or HPV-18
Description: as for outcome 4
Time Frame: Up to year 7
Population: as for outcome 32
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 171 | 145
Subjects
  HPV-16/18 (N=171;139) | 0 | 0
  HPV-16 (N=171;144) | 0 | 0
  HPV-18 (N=171;145) | 0 | 0

63. Secondary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With Any Oncogenic HPV Type
Description: as for outcome 5
Time Frame: Up to year 7
Population: as for outcome 35
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 157 | 138
Subjects
  Including HPV-16 or 18 (N=157;137) | 5 | 4
  Without HPV-16 or 18 (N=157;138) | 5 | 4

64. Secondary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With Individual Oncogenic Non-vaccine HPV Types
Description: as for outcome 6
Time Frame: Up to year 7
Population: as for outcome 35
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 195 | 177
Subjects
  HPV-31 (N= 193; 173) | 0 | 2
  HPV-33 (N=191; 175) | 0 | 0
  HPV-35 (N=192; 173) | 1 | 1
  HPV-39 (N=191; 168) | 0 | 1
  HPV-45 (N=195; 177) | 1 | 0
  HPV-51 (N=183; 167) | 2 | 0
  HPV-52 (N=177; 160) | 2 | 1
  HPV-56 (N=189; 175) | 0 | 0
  HPV-58 (N=188; 174) | 1 | 1
  HPV-59 (N=195; 177) | 0 | 0
  HPV-66 (N=183; 164) | 0 | 1
  HPV-68 (N=191; 174) | 1 | 0

65. Secondary Outcome: Number of Subjects With Persistent Infection (12-month Definition) With HPV-16 and/or HPV-18
Description: as for outcome 7
Time Frame: Up to year 7
Population: as for outcome 35
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 171 | 150
Subjects
  HPV-16/18 (N=171;146) | 0 | 0
  HPV-16 (N=171;148) | 0 | 0
  HPV-18 (N=171;150) | 0 | 0

66. Secondary Outcome: Number of Subjects With Persistent Infection (12-month Definition) With Any Oncogenic HPV Type
Description: as for outcome 8
Time Frame: Up to year 7
Population: as for outcome 35
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 158 | 138
Subjects
  Including HPV-16 or 18 (N=158;138) | 0 | 0
  Without HPV-16 or 18 (N=158;138) | 0 | 0

67. Secondary Outcome: Number of Subjects With Persistent Infection (12-month Definition) With Individual Oncogenic Non-vaccine HPV Types
Description: as for outcome 9
Time Frame: Up to year 7
Population: as for outcome 35
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 196 | 179
Subjects
  HPV-31 (N=194;174) | 0 | 0
  HPV-33 (N=194;177) | 0 | 0
  HPV-35 (N=192;178) | 0 | 0
  HPV-39 (N=192;173) | 0 | 0
  HPV-45 (N=196;179) | 0 | 0
  HPV-51 (N=190;175) | 0 | 0
  HPV-52 (N=183;166) | 0 | 0
  HPV-56 (N=193;178) | 0 | 0
  HPV-58 (N=193;178) | 0 | 0
  HPV-59 (N=196;179) | 0 | 0
  HPV-66 (N=187;170) | 0 | 0
  HPV-68 (N=192;177) | 0 | 0

68. Secondary Outcome: Number of Subjects With Histopathologically-confirmed CIN1+ Associated With HPV-16 or HPV-18 Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: CIN1+ was defined as CIN grades 1,2 and 3, adenocarcinoma in situ (AIS) and invasive cervical cancer.
  Subjects with an event did not report the same event in the earlier studies. Subjects were DNA negative for the 14 oncogenic HPV types and had normal cytology at baseline in the primary study. Subjects with an event were DNA negative for the corresponding HPV type at Month 6 in the primary study.
Time Frame: Up to year 7
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 191 | 178
Subjects
  HPV-16/18 (N=191;175) | 0 | 0
  HPV-16 (N=191;176) | 0 | 0
  HPV-18 (N=191;178) | 0 | 0

69. Secondary Outcome: Number of Subjects With Histopathologically Confirmed CIN1+ Associated With Oncogenic HPV Types Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: as for outcome 11
Time Frame: Up to year 7
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 191 | 179
Subjects
  Including HPV-16 or 18 (N=191;179) | 0 | 0
  Without HPV-16 or 18 (N=191;179) | 0 | 0

70. Secondary Outcome: Number of Subjects With Histopathologically Confirmed CIN1+ Associated With Individual Oncogenic Non-Vaccine HPV Types Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: as for outcome 12
Time Frame: Up to year 7
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 214 | 201
Subjects
  HPV-31 (N=213;199) | 0 | 0
  HPV-33 (N=212;199) | 0 | 0
  HPV-35 (N=211;198) | 0 | 0
  HPV-39 (N=214;201) | 0 | 0
  HPV-45 (N=213;200) | 0 | 0
  HPV-51 (N=207;198) | 0 | 0
  HPV-52 (N=210;196) | 0 | 1
  HPV-56 (N=211;201) | 0 | 0
  HPV-58 (N=213;198) | 0 | 0
  HPV-59 (N=212;200) | 0 | 0
  HPV-66 (N=211;195) | 0 | 0
  HPV-68 (N=213;201) | 0 | 0

71. Secondary Outcome: Number of Subjects With Histopathologically-confirmed CIN2+ Associated With HPV-16 or HPV-18 Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: as for outcome 13
Time Frame: Up to year 7
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 191 | 178
Subjects
  HVP-16/18 (N=191;176) | 0 | 0
  HPV-16 (N=191;177) | 0 | 0
  HPV-18 (N=191;178) | 0 | 0

72. Secondary Outcome: Number of Subjects With Histopathologically Confirmed CIN2+ Associated With Oncogenic HPV Types Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: as for outcome 14
Time Frame: Up to year 7
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 191 | 179
Subjects
  Including HPV-16 or 18 (N=191;179) | 0 | 0
  Without HPV-16 or 18 (N=191;179) | 0 | 0

73. Secondary Outcome: Number of Subjects With Histopathologically Confirmed CIN2+ Associated With Individual Oncogenic Non-Vaccine HPV Types Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: as for outcome 45
Time Frame: Up to year 7
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 214 | 201
Subjects
  HPV-31 (N=213;200) | 0 | 0
  HPV-33 (N=212;200) | 0 | 0
  HPV-35 (N=212;198) | 0 | 0
  HPV-39 (N=214;201) | 0 | 0
  HPV-45 (N=213;200) | 0 | 0
  HPV-51 (N=209;199) | 0 | 0
  HPV-52 (N=210;198) | 0 | 1
  HPV-56 (N=211;201) | 0 | 0
  HPV-58 (N=213;199) | 0 | 0
  HPV-59 (N=212;200) | 0 | 0
  HPV-66 (N=212;197) | 0 | 0
  HPV-68 (N=213;201) | 0 | 0

74. Secondary Outcome: Number of Subjects With Abnormal Cytology Greater Than or Equal to Atypical Squamous Cells of Undetermined Significance (ASC-US) Associated With an HPV 16 and/or HPV-18 Cervical Infection
Description: as for outcome 16
Time Frame: Up to year 7
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 191 | 169
Subjects
  HPV-16/18 (N=190;158) | 0 | 0
  HPV-16 (N=190;164) | 0 | 0
  HPV-18 (N=191;169) | 0 | 0

75. Secondary Outcome: Number of Subjects With Abnormal Cytology Greater Than or Equal to Atypical Squamous Cells of Undetermined Significance (ASC-US) Associated With Oncogenic HPV Types Cervical Infection
Description: as for outcome 17
Time Frame: Up to year 7
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 188 | 176
Subjects
  Including HPV-16 or 18 (N=188;175) | 3 | 8
  Without HPV-16 or 18 (N=188;176) | 3 | 8

76. Secondary Outcome: Number of Subjects With Abnormal Cytology Greater Than or Equal to Atypical Squamous Cells of Undetermined Significance (ASC-US) Associated With Individual Oncogenic Non-vaccine HPV Types Cervical Infection
Description: as for outcome 18
Time Frame: Up to year 7
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 212 | 198
Subjects
  HPV-31 (N=209;192) | 0 | 1
  HPV-33 (N=210;194) | 0 | 0
  HPV-35 (N=209;194) | 0 | 1
  HPV-39 (N=209;189) | 0 | 1
  HPV-45 (N=212;196) | 1 | 0
  HPV-51 (N=194;187) | 0 | 1
  HPV-52 (N=197;176) | 1 | 2
  HPV-56 (N=200;194) | 0 | 0
  HPV-58 (N=206;191) | 0 | 1
  HPV-59 (N=209;198) | 0 | 1
  HPV-66 (N=206;186) | 1 | 1
  HPV-68 (N=210;194) | 1 | 0

77. Secondary Outcome: Number of Subjects With Abnormal Cytology Greater Than or Equal to Low-grade Squamous Intraepithelial Lesion (LSIL) Associated With an HPV 16 and/or HPV-18 Cervical Infection
Description: as for outcome 19
Time Frame: Up to year 7
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 191 | 175
Subjects
  HPV-16/18 (N=190;167) | 0 | 0
  HPV-16 (N=190;170) | 0 | 0
  HPV-18 (N=191;175) | 0 | 0

78. Secondary Outcome: Number of Subjects With Abnormal Cytology Greater Than or Equal to Low-grade Squamous Intraepithelial Lesion (LSIL) Associated With Oncogenic HPV Types Cervical Infection
Description: as for outcome 17
Time Frame: Up to year 7
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 189 | 178
Subjects
  Including HPV-16 or 18 (N=189;178) | 2 | 6
  Without HPV-16 or 18 (N=189;178) | 2 | 6

79. Secondary Outcome: Number of Subjects With Abnormal Cytology Greater Than or Equal to Low-grade Squamous Intraepithelial Lesion (LSIL) Associated With Individual Oncogenic Non-vaccine HPV Types Cervical Infection
Description: as for outcome 18
Time Frame: Up to year 7
Population: as for outcome 40
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 212 | 199
Subjects
  HPV-31 (N=210;194) | 0 | 1
  HPV-33 (N=211;197) | 0 | 0
  HPV-35 (N=209;196) | 0 | 0
  HPV-39 (N=211;192) | 0 | 1
  HPV-45 (N=212;197) | 1 | 0
  HPV-51 (N=203;190) | 0 | 1
  HPV-52 (N=202;184) | 0 | 2
  HPV-56 (204;194) | 0 | 0
  HPV-58 (N=209;195) | 0 | 0
  HPV-59 (N=212;199) | 0 | 1
  HPV-66 (N=209;187) | 0 | 1
  HPV-68 (N=211;198) | 1 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events: during the follow-up period up to Year 9.
Description: Only serious adverse events were assessed in the study and no other symptoms.
Arm/Group | Cervarix Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 20/224 | 11/213
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=224) | Placebo Group (N=213)
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 5 | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 2 | 2
Appendicitis (Infections and infestations) | 2 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 1 | 0
Benign hydatidiform mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Bronchiectasis (Infections and infestations) | 1 | 0
Depression suicidal (Psychiatric disorders) | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Gestational diabetes (Metabolism and nutrition disorders) | 1 | 0
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Myelitis (Nervous system disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Renal artery thrombosis (Renal and urinary disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Varicose vein (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Interim analysis at Year 7 and Year 8 are superseded by the final analysis at Year 9.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.